CLINICAL TRIAL: NCT03091296
Title: Diurnal Testosterone Concentrations in Men With and Without Testosterone Deficiency
Brief Title: Diurnal Testosterone Concentration
Status: Completed | Type: Observational
Sponsor: Men's Health Boston (Other)
Responsible Party: Principal Investigator, Dr. Abraham Morgentaler, Director, Men's Health Boston
Other Study IDs: MHB022
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Testosterone Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men with testosterone deficiency: Screening testosterone concentration of less than 350 ng/dL
- Men without testosterone deficiency: Screening testosterone concentration of greater than 350 ng/dL

SUMMARY:
In this case-controlled, observational study, 24 subjects will participate in a 12-hour blood collection with a single blood draw at +24 hours. 12 men will have low testosterone levels (hypogonadism) and 12 men will have normal testosterone levels. Blood samples will be drawn every 2 hours and later analyzed for total testosterone and calculated free testosterone. The primary objective of this study is to assess the degree of diurnal variation in men with testosterone deficiency.

ELIGIBILITY:
Inclusion Criteria:

Men with testosterone deficiency:

* Ability to read, write, and understand English
* Male sex at birth
* Age greater than or equal to 18
* Age less than 46
* Diagnosed with testosterone deficiency prior to visit 1
* Screening testosterone concentration of less than 350 ng/dL
* Willing and able to comply with the study protocol
* Willing to provide informed consent for this study
* No previous exposure to exogenous T unless off therapy for at least 4 weeks

Men without testosterone deficiency:

* Ability to read, write, and understand English
* Male sex at birth
* Age greater than or equal to 18
* Age less than 46
* Never diagnosed with testosterone deficiency
* Screening testosterone concentration of greater than 350 ng/dL
* Willing and able to comply with the study protocol
* Willing to provide informed consent for this study
* No previous exposure to exogenous T

Exclusion Criteria:

* Previous exposure to exogenous T, clomiphene citrate, or other Selective Estrogen Receptor Modulators, unless off therapy for at least 4 weeks
* Serious psychiatric disease or uncontrolled medical illness, as suspected from the history or clinical examination
* Used any sex hormones or steroidal anabolic drug supplements within 28 days before screening testosterone collection
* Incapable of giving informed consent or complying with the protocol

Ages: 18 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 male subjects (12 with TD and 12 without TD)
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Change in levels of serum total testosterone concentration | 24 hours
  Blood samples analyzed by Beckman assays and equipment
Change in levels of serum calculated free testosterone concentration | 24 hours
  Blood samples analyzed by Beckman assays and equipment

SECONDARY OUTCOMES:
Change in levels of estradiol | 24 hours
  Blood samples analyzed by Beckman assays and equipment
Change in levels of serum LH | 24 hours
  Blood samples analyzed by Beckman assays and equipment
Change in levels of serum FSH | 24 hours
  Blood samples analyzed by Beckman assays and equipment
Change in levels of serum SHBG | 24 hours
  Blood samples analyzed by Beckman assays and equipment
Change in levels of whole blood hematocrit | 24 hours
  Blood samples analyzed by Quest assays and equipment

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Morgentaler, MD, Principal Investigator — Men's Health Boston, Harvard Medical School
Locations (1):
- Men's Health Boston, Chestnut Hill, Massachusetts, United States